CLINICAL TRIAL: NCT00682669
Title: Asthma and Mindfulness-Based Stress Reduction (MBSR)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002938 (NIH)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: Asthma; Mindfulness-based stress reduction; Peak expiratory flow rate; Spirometry; Quality of life
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBSR (Experimental): A mindfulness-based stress reduction (MBSR) program consisting of an 8-week, 9-session intervention based on systematic and intensive training in mindfulness meditation and mindful hatha yoga and their application to every day life.
  Interventions: Behavioral: MBSR
- HLC (Active Comparator): A Healthy Living Course (HLC) consisting of an 8-week program of lectures and discussion on health-related topics.
  Interventions: Behavioral: HLC

INTERVENTIONS:
Behavioral: MBSR — A mindfulness-based stress reduction (MBSR) program consisting of an 8-week, 9-session intervention based on systematic and intensive training in mindfulness meditation and mindful hatha yoga and their application to every day life.
  Arms: MBSR
Behavioral: HLC — An 8-week program consisting of lectures and discussion of health-related topics.
  Arms: HLC

SUMMARY:
Asthma is one of the four most common chronic disorders in adults, affecting 14 million adults in the United States and costing an estimated 7.9 billion dollars in medical care and 5.3 billion dollars in lost work or school. About 40% of asthmatics report using some form of complementary and alternative medicine approach to help reduce their asthma symptoms, but there is little evidence for their effectiveness. Mindfulness-based stress reduction (MBSR) is a group based program shown to reduce medical symptoms and improve quality of life for patients with many different chronic diseases. The goals of the proposed randomized controlled trial are to collect preliminary data on the effect of MBSR on quality of life, symptoms, and lung function in mild and moderate-severity asthmatics and to refine recruitment and data collection procedures for a future, larger clinical trial.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory disease that affects 7% or 14 million adults in the United States. It is one of the four most common chronic disorders in adults, costing an estimated 7.9 billion dollars in medical care and 5.3 billion dollars in lost work or school. Approximately 40% of asthmatics report using some form of complementary and alternative medicine (CAM) approach to help alleviate their asthma symptoms, but there is little evidence for their effectiveness. Breathing and relaxation techniques, including yoga appear most promising. Mindfulness-based stress reduction (MBSR) is a group-based program developed at the University of Massachusetts Medical School (UMMS) that focuses on the cultivation of mindfulness through formal meditation practices and the integration of mindfulness into everyday life as a coping resource to deal with physical symptoms, chronic medical conditions, and difficult emotional situations. MBSR has been shown to be an effective adjunctive intervention in reducing medical symptoms for a broad range of stress-related disorders and chronic diseases, reducing psychological distress anxiety and depression, and improving quality of life. A small preliminary study conducted by our research team found improvements in measures of quality of life, locus of control, stress, and anxiety immediately following the completion of the MBSR program.

The overall goal of the proposed two year exploratory study is to conduct a randomized controlled trial (RCT) to test and optimize recruitment and data collection procedures and to collect preliminary data on the effect of MBSR on behavioral and psychological aspects of asthma and lung function to support justification for a larger clinical trial should the results of this study be promising. Eighty-two adults ages 21 and older with a physician-documented diagnosis of asthma classified as either mild or moderate documented will be recruited for seventy participants at final follow-up. Participants will be randomly assigned to one of two conditions stratified by asthma severity: (1) MBSR, or (2) Healthy Living Course (HLC) attention control condition. Participant assessments will occur at study entry (baseline) and at 10-week, 6- and 12-month follow-up. The primary aim of the project is to evaluate the efficacy of the MBSR program in improving quality of life and lung function as assessed by change from baseline to two-week average morning peak expiratory flow (PEF) compared to HLC participants. Secondary aims are to evaluate the effect of the MBSR program on reducing asthma rescue medication use, frequency of asthma exacerbations (prednisone therapy), asthma symptoms, healthcare utilization, number of days of work or school missed, peak expiratory flow (PEF) variation, and psychological distress, and in improving asthma control, asthma-related internal locus of control, and lung function as assessed by spirometry (FEV1).

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of asthma from their physician
* meet criteria for mild persistent or moderate persistent asthma
* able to read and understand English
* able to complete informed consent process and study data collection procedures
* 21 or older

Exclusion Criteria:

* current smoker
* other lung diseases besides asthma
* cancer, except non-melanoma skin cancer
* currently receiving treatment for symptomatic cardiovascular disease
* on psychotropic medications in the prior 6 months
* psychiatric hospitalization in the last 2 years
* has taken the MBSR program in the past
* currently practicing meditation or yoga on a regular basis

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Quality of life and lung function. | 10 week, 6- and 12-month post baseline

SECONDARY OUTCOMES:
Reduce asthma symptoms, exacerbations and health care utilization | 10-week, 6- and 12-month post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Pbert L, Madison JM, Druker S, Olendzki N, Magner R, Reed G, Allison J, Carmody J. Effect of mindfulness training on asthma quality of life and lung function: a randomised controlled trial. Thorax. 2012 Sep;67(9):769-76. doi: 10.1136/thoraxjnl-2011-200253. Epub 2012 Apr 27. PMID 22544892